CLINICAL TRIAL: NCT05313269
Title: Inter-fascial Plane Between the SArtorius Muscle and FEmoral Artery (ISAFE): a Novel Technique for Adductor Canal Catheter Insertion.
Brief Title: Inter-fascial Plane Between the SArtorius Muscle and FEmoral Artery (ISAFE)
Acronym: ISAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Hermann dos Santos Fernandes, Principal Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-0258-A
Record Dates: First submitted 2022-03-28; First posted 2022-04-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Anesthesia, Conduction; Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ISAFE technique (Experimental): Adductor canal block catheter tip located in the fascial plane between sartorious muscle and femoral artery.
  Interventions: Other: ISAFE technique for adductor canal catheter insertion
- Conventional technique (Active Comparator): Adductor canal block catheter tip located in lateral to the femoral artery.
  Interventions: Other: Conventional technique for adductor canal catheter insertion

INTERVENTIONS:
Other: ISAFE technique for adductor canal catheter insertion — Adductor canal block catheter tip located in the fascial plane between sartorious muscle and femoral artery.
  Other Names: ISAFE approach
  Arms: ISAFE technique
Other: Conventional technique for adductor canal catheter insertion — Adductor canal block catheter tip located lateral to the femoral artery.
  Other Names: Conventional approach
  Arms: Conventional technique

SUMMARY:
Total knee arthroplasty (TKA) is a frequent performed surgery. Adequate pain management is an important feature. Analgesic duration of single shot nerve blocks is limited to no more than 24h. Conversely, the use of continuous nerve block (CNB) through a perineural catheter and infusion of local anesthetic may increase duration of analgesia and provide better outcomes. Continuous adductor canal block (CACB) has been proven superior when compared to single-injection adductor canal block (SACB) for TKA analgesia. However, safety concerns such as intravenous insertion, nerve injury, or catheter displacement must always be considered. The purpose of this study is to evaluate the Inter-fascial Plane between SArtorius Muscle and FEmoral Artery (ISAFE) approach for adductor canal catheter placement, in terms of catheter dislodgment, clinical effectiveness and complications, in comparison with the classical approach, as TKA postoperative analgesia modality. We hypothesize that ISAFE approach can result in a smaller rate of dislodgments in the way that it increases the clinical benefit of CACB.

DETAILED DESCRIPTION:
Introduction Total knee arthroplasty (TKA) is an effective treatment for end stage osteoarthritis, with over 75,000 TKA performed in Canada annually (https://www.cihi.ca/en/hip-and-knee-replacements-in-canada-cjrr-annual-report) and an incidence rate of 135 per 100000 of population, among OECD countries, in 2017 (https://www.oecd-ilibrary.org/sites/2fc83b9a-en/index.html?itemId=/content/component/2fc83b9a-en). Historically, TKA has been associated with a significant level of postoperative pain, which can be a barrier to an early discharge. In order to optimize analgesia and minimize opioid consumption and its associated side effects, regional anesthesia techniques traditionally used for TKA include peripheral nerve blocks such as femoral and adductor canal blocks (ACB). These blocks typically provide superior analgesia by anesthetizing peripheral nerves that supply sensory innervation to the surgical site. Specifically, the ACB is of great value as it does not cause the quadriceps weakness motor block that the femoral nerve block provides, thereby facilitating early patient mobilization and discharge. An even newer technique has also emerged called the IPACK (infiltration between the popliteal artery and capsule of the knee), which has been used in some centers to replace sciatic blocks to cover posterior knee pain experienced by many TKA patients, without affecting motor function of the lower leg and foot. Recently, continuous adductor canal blocks (CACB) via an inserted adductor canal catheter (ACC) have started to replace single injection blocks, as they extend the block duration and offer prolonged analgesia. Studies evaluating CACB have it to be superior when compared to single-injection adductor canal block (SACB) for inpatients post-TKA analgesia. Currently at Sinai Health, CACB has become the standard of care for inpatient TKA with all patients routinely being offered this analgesic modality.

Placing a successful ACC is not without risk or technical difficulty. The classic insertion approach involves placing the tip of the ACC near the saphenous nerve in the mid-thigh area. The proximity of the femoral artery (FA) and femoral vein (FV) to the saphenous nerve adds the risk of vascular puncture and intravascular placement of the ACC. Specifically, the FV is deeper and more difficult to visualize as it is compressible, and can be easily punctured if the needle is manipulated in its proximity. Intravenous placement of an ACC will result local anesthetic systemic toxicity (LAST), a potentially lethal albeit very rare complication, and therefore effort should be made to avoid this at all costs. Lastly, a more common obstacle when placing ACC is ensuring that the catheter stays inside the adductor canal. Since the adductor canal itself is very narrow, the catheter tip can easily migrate out of the canal with patient movement and mobilization, resulting in no sensory block and inadequate analgesia. It is not uncommon for patients to initially have well working CACB, but to experience significant rebound pain on postoperative days (POD) 1 or 2 due to catheter dislodgement out of the canal.

In order to address these issues we have developed a novel insertion approach for ACC is inserted into the inter-fascial plane between the Sartorius muscle and femoral artery (ISAFE). In this technique, the needle is inserted into the plane between the sartorius muscle and FA. A catheter is then threaded between the artery and muscle, well away from the FV. This facilitates keeping the needle away from the vein and maintaining more catheter length inside the adductor canal, thereby preventing catheter dislodgement. The insertion angle of the needle is shallower when compared to the classic ACC technique, allowing for better needle visualization, and steering clear of the FV. While the needle is still in close proximity to the FA, this vessel is easier to visualize, more difficult to puncture, and is much less likely to result in LAST.

While the ISAFE technique is an exciting novel approach for ACC insertion, it still requires evaluation in terms of analgesia efficacy and superiority in terms of reducing catheter dislodgement.

Significance There are no published prospective randomized controlled trials that compare insertion techniques for ACC and their respective outcomes in terms of catheter positioning, dislodgement, and safety. As TKA is a frequent type of surgery and has the prediction to increase its incidence for the next years, there is significant importance in investigations about interventions which may improve its recovery in an outpatient regime. A postoperative analgesic technique that offers better pain control, has less adverse effects, reduces the opioid analgesia requirement and is safe may have additional impact on decreasing health care cost and may lead to an enhanced recovery and better quality of life.

Objectives The primary objective will be to evaluate the rate of ACC dislodgement when using the ISAFE approach for CACB in patients undergoing TKA (by measuring cumulative postoperative opioid consumption), in comparison with the classical ACC insertion technique.

The secondary objective is to assess the quality of analgesia as measured by pain scores and opioid consumption, and complications relating to the perineural catheter use.

Hypothesis The ISAFE insertion approach for ACC in patients undergoing TKA will lead to a reducing in catheter dislodgement rates.

Methods Study type This will be a Randomized controlled prospective trial, blinded for patient and evaluator, in patients undergoing inpatient TKA at Sinai Health. After Hospital's Ethics in Research Board approval, the recruitment will begin. Patients will be assessed about their eligibility for participating and after plain clear information about the study interventions they will or will not authorize their inclusion and data collection, through the signature of a written consent.

Perioperative management and interventions The subjects will have their surgeries booked in advance and they will be submitted to the pre anesthesia consult at the Pre Admission Unit a few days before the surgery. The study proposal will be explained to the patients on that occasion and they will receive a booklet with the information about the study as well as the consent form that they will bring home to review. They will have the time between the pre anesthesia assessment and the surgery (at least 24 hours) to review and consent to the study.

Patients will be randomized to one of the two groups using a computer-generated random numbers table. The randomization will be done before the beginning of the study and will define which study number is going to be managed as intervention group (ISAFE approach) or control group (classic approach). Each patient will receive a study number following the order of their entrance on the study and that number will be already linked for one of the two groups. Closed envelopes will be prepared ahead and each of them will have the name of the group related to its study number. Once the the patient is included, the professional who inserts the catheter will check inside the envelope which group the patient is randomized to, in order to perform the predicted technique. A list with the study numbers and the randomization will be kept by the research assistant, under password protection, and will be shared with other researches only after recruitment is finished. The research coordinator, and the professional who performs the postoperative adductor canal assessments will be blinded to which group each patient was randomized to. The professional who inserts the catheters will not be blinded as they will need to know which insertion approach to take.

All patients will receive the same perioperative management. Patients will initially be brought to a dedicated block room where a safety checklist will be performed by the block room team. Standard Canadian Anesthesia Society monitoring will be provided. Mild sedation with Midazolam 0.5-2mg and Fentanyl 25-100mcg might be administered for anxiolysis and analgesia. After proper cleaning of the ipsilateral thigh, under sterile technique and ultrasound guidance (Sonosite Edge II ultrasound machine), an adductor canal block (injection of 15 mL of Ropivacaine 0.5% with epinephrine 1:200,000) and an IPACK block (injection of 15 mL of Ropivacaine 0.25% with epinephrine 1:200,000) will be performed. Cumulative local anesthetic doses will be preemptively calculated to avoid a total Ropivacaine dose of > 3mg/kg. After the peripheral nerve blocks, all patients will receive standard spinal or general anesthesia. All intraoperative opioids administered will be recorded. In the intra-operative period, each patient will receive IV Cefazolin 2g, Tranexamic acid 20mg/kg, Dexamethasone 0.1mg/kg, and Ondansetron 4mg. At the end of the procedure the surgeons will infiltrate the surgical site with 200 mg of Ropivacaine 0.2%.

After surgery, the patient will be taken to the Post Anesthesia Care Unit. At this moment, an Arrow® (StimuCath® Continuous Peripheral Nerve Block Catheter) continuous adductor canal block catheter will be inserted using a Sonosite Edge II ultrasound machine. A bolus of 5-10mL of saline solution (NaCl 0.9%) with epinephrine 1:200,000 will be given, after negative aspiration, following adductor canal catheter insertion and the patient will be monitored for any heart rate change in order to rule out intravascular catheter placement. The catheter will be well secured with an adhesive fixation device to avoid displacement. Following catheter placement, the catheter will be aspirated to check for blood to ensure there is no intravascular placement. The peripheral nerve catheter will be connected to an elastomeric infusion pump and will infuse Ropivacaine 0.2% at a rate of 5 ml/hour, as per the standard Sinai Health practice for inpatient CACB. Adductor canal catheter will be placed following the surgery in the post-anesthetic care unit in order to avoid catheter displacement by the thigh tourniquet used intraoperatively. The adductor canal catheter stays in place infusing for 48 hours. The patients are discharged home after achieving the discharge criteria by orthopedics team in charge, keeping the peripheral nerve catheter with the same infusion rate, if they go home before completing the 48 hours of infusion. Prior to going home, patients receive education and written information (educational pamphlet) regarding monitoring for local anesthetic systemic toxicity symptoms, possible CABC associated complications including potential transient muscle weakness, and instructions on patient removal of the catheter after infusion end. This pamphlet contains contact information for anesthesia team or Acute Pain Service, in case of any events, adverse effects or questions the patients may have about the peripheral nerve catheter. A phone number to contact each patient at home is collected before they are discharged and they are followed up by phone calls, during the infusion period. This is already done as standard of care for all knee arthroplasty surgeries.Standard oral analgesic scheme will be prescribed to every patient (Acetaminophen 650mg QID, Celecoxib 200mg BID, Hydromorphone 1-2mg PRN Q4Hs).

Sample size The sample size was calculated based on previous study that ACC dislodgement rate of 13%. This study measured catheter dislodgement at the skin, so we believe this rate significantly underestimates the rate of dislodgement out of the adductor canal and that sonographic assessments will have a much higher sensitivity for such events. Local pilot data suggests that using the ISAFE approach, ACC dislodgements are only 5%. Using a predicted catheter dislodgement rate of 25% for conventional approach, and an expected reduction for of dislodgement rate down to 5% with ISAFE approach, considering α=0.05 and a power of 80%, 49 subjects will be needed in each group for a total of 98 patients. To compensate for anticipated dropouts from the study, we plan for an inclusion of 100 patients.

Study data analysis Normal distributed variables values will be presented and analyzed as mean values +- standard deviation. Non-normal distributed variables values will be presented and analyzed as median and minimum and maximum values. Qualitative variables will be presented as frequency of occurrence. Statistical test to be performed might be: t-Student, Kruskal-Wallis and Chi-square. Statistical software will be used for analysis: SPSS 13.0 for Windows (SPSS Inc, Chicago, IL, USA) and GraphPad Prism Version 4.00 for Windows (GraphPad Software, San Diego, CA, USA).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary or revision Total Knee Arthroplasty in the inpatient setting. Non-pregnant patients older than 21 years of age, with American Society of Anesthesiologists (ASA) physical status I-IV.

Exclusion Criteria:

* Patients undergoing outpatient TKA. Chronic opioid use of oral morphine 30mg equivalent per day for last 2 consecutive weeks. Patients with contraindications to the insertion of an adductor canal catheter (severe anatomic abnormalities, local or systemic infection, or a history of previous surgery at the site of catheter placement).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Catheter dislodgement | 24 hours
  Rate of migration of the catheter tip to outside the adductor canal, verified by ultrasound assessment

SECONDARY OUTCOMES:
Pain intensity | 24 and 48 hours
  Numerical verbal scale for pain intensity (from 0 to 10, 0 being no pain and 10 the worst pain ever)
Opioid consumption | 24 and 48 hours
  Amount of opioid in Oral Morphine Equivalents
Number of attempts for catheter insertion | 4 hours
  Number of attempts that were necessary for adductor canal catheter insertion
Incidence of catheter insertion related complications | 4 hours
  Paresthesia, catheter leakage, blood aspiration or vascular puncture
Potential complications related to continuous adductor canal block catheter | 24 and 48 hours
  Patients are asked about ipsilateral lower limb weakness (any degree of weakness), falls, signs of local infection (redness, pain, swelling and yellow exudate), pruritus, burning, tingling and shock sensation on saphenous nerve territory, symptoms of local anesthetic systemic toxicity (numbness on lips or tongue, metal taste, tinnitus), leakage from catheter or insertion site, and catheter exteriorization
Ultrasound assessment of the dislodgement of the catheter | 24 hours
  Distance between the catheter location and its original position and its distance from the saphenous nerve
Incidence of sensory block | 24 hours
  Block to ice sensation on saphenous nerve territory

CONTACTS AND LOCATIONS:
Overall Officials: Yehoshua Gleicher, MD, MSc, Study Chair — University of Toronto
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized REDCap data base, after conclusion of the study.
Supporting Information: Study Protocol, CSR
Time Frame: At the conclusion of the study

REFERENCES:
- [Background] Price AJ, Alvand A, Troelsen A, Katz JN, Hooper G, Gray A, Carr A, Beard D. Knee replacement. Lancet. 2018 Nov 3;392(10158):1672-1682. doi: 10.1016/S0140-6736(18)32344-4. PMID 30496082
- [Background] Cullom C, Weed JT. Anesthetic and Analgesic Management for Outpatient Knee Arthroplasty. Curr Pain Headache Rep. 2017 May;21(5):23. doi: 10.1007/s11916-017-0623-y. PMID 28283810
- [Background] Sankineani SR, Reddy ARC, Eachempati KK, Jangale A, Gurava Reddy AV. Comparison of adductor canal block and IPACK block (interspace between the popliteal artery and the capsule of the posterior knee) with adductor canal block alone after total knee arthroplasty: a prospective control trial on pain and knee function in immediate postoperative period. Eur J Orthop Surg Traumatol. 2018 Oct;28(7):1391-1395. doi: 10.1007/s00590-018-2218-7. Epub 2018 May 2. PMID 29721648
- [Background] Yu R, Wang H, Zhuo Y, Liu D, Wu C, Zhang Y. Continuous adductor canal block provides better performance after total knee arthroplasty compared with the single-shot adductor canal block?: An updated meta-analysis of randomized controlled trials. Medicine (Baltimore). 2020 Oct 23;99(43):e22762. doi: 10.1097/MD.0000000000022762. PMID 33120783
- [Background] Leung P, Dickerson DM, Denduluri SK, Mohammed MK, Lu M, Anitescu M, Luu HH. Postoperative continuous adductor canal block for total knee arthroplasty improves pain and functional recovery: A randomized controlled clinical trial. J Clin Anesth. 2018 Sep;49:46-52. doi: 10.1016/j.jclinane.2018.06.004. Epub 2018 Jun 8. PMID 29890381
- [Background] Edwards RM, Currigan DA, Bradbeer S, Mitchell C. Does a catheter over needle system reduce infusate leak in continuous peripheral nerve blockade: a randomised controlled trial. Anaesth Intensive Care. 2018 Sep;46(5):468-473. doi: 10.1177/0310057X1804600507. PMID 30189820
- [Background] Dos Santos Fernandes H, Siddiqui N, Peacock S, Vidal E, Wolfstadt J, Gleicher Y. Inter-fascial space between SArtorius muscle and FEmoral artery (ISAFE): A suggested approach for Adductor Canal catheter placement. J Clin Anesth. 2022 Feb;76:110571. doi: 10.1016/j.jclinane.2021.110571. Epub 2021 Nov 8. No abstract available. PMID 34763273
- [Background] Sun C, Zhang X, Song F, Zhao Z, Du R, Wu S, Ma Q, Cai X. Is continuous catheter adductor canal block better than single-shot canal adductor canal block in primary total knee arthroplasty?: A GRADE analysis of the evidence through a systematic review and meta-analysis. Medicine (Baltimore). 2020 May;99(20):e20320. doi: 10.1097/MD.0000000000020320. PMID 32443383